CLINICAL TRIAL: NCT07017699
Title: The Deucravacitinib Pregnancy Exposure Study: A Prospective Observational Study of Deucravacitinib Safety in Pregnancy
Brief Title: A Study to Assess Deucravacitinib Safety in Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-1111
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis (PsO)
Keywords: Psoriasis (PsO)
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Deucravacitinib Cohort: Pregnant participants with psoriasis exposed to deucravacitinib treatment
  Interventions: Drug: Deucravacitinib
- Other Systemic Treatment Cohort: Pregnant participants with psoriasis exposed to other systemic treatments for PsO
  Interventions: Drug: Other systemic treatments for PsO
- Unexposed Cohort: Pregnant participants without psoriasis or any other autoimmune diseases

INTERVENTIONS:
Drug: Deucravacitinib — According to product label
  Groups: Deucravacitinib Cohort
Drug: Other systemic treatments for PsO — According to product label
  Groups: Other Systemic Treatment Cohort

SUMMARY:
The purpose of this study is to assess pregnancy and infant outcomes among pregnant participants enrolled in an established North American pregnancy registry (Organization of Teratology Information Specialists [OTIS]) who were exposed to deucravacitinib.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: Deucravacitinib-exposed cohort

* Currently pregnant during the enrollment period
* Diagnosed with psoriasis (PsO) validated by medical records when possible
* Exposure to deucravacitinib for any number of days, at any dose, and at any time from 2 days prior to date of conception (DOC) to the end of pregnancy
* Agree to the conditions and requirements of the study including the interview schedule, release of medical records, and the dysmorphology examination of live born infants

Cohort 2: PsO Disease-matched unexposed comparator cohort

* Currently pregnant during the enrollment period
* Diagnosed with PsO validated by medical records when possible
* May be exposed to systemic treatments for PsO
* Agree to the conditions and requirements of the study including the interview schedule, release of medical records, and the dysmorphology examination of live born infants

Cohort 3: Non-disease unexposed comparator cohort

* Currently pregnant during the enrollment period
* Agree to the conditions and requirements of the study including the interview schedule, release of medical records, and the dysmorphology examination of live born infants

Exclusion Criteria

Cohort 1: Deucravacitinib-exposed cohort

* Pregnant women who have enrolled in this cohort study with a previous pregnancy
* Pregnant women who have used deucravacitinib for an indication other than PsO
* Women who do not have exposure to deucravacitinib anytime from 2 days prior to DOC to the end of pregnancy
* Women who have exposure to another oral tyrosine kinase 2 (TYK2) inhibitor or any oral Janus kinase (JAK) inhibitor from within 5 half-lives of DOC to the end of pregnancy
* Women who have exposure to methotrexate or an oral retinoid
* Retrospective enrollment after the outcome of pregnancy is known (ie, the pregnancy has ended prior to enrollment)
* Results of a diagnostic test are positive for an major congenital malformation(s) (MCM) prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate an MCM

Cohort 2: Disease-matched unexposed comparator cohort

* Pregnant women who have enrolled in this cohort study with a previous pregnancy
* Women who have exposure to deucravacitinib or any other oral TYK2 inhibitor except deucravacitinib, or any oral JAK inhibitor from within 5 half-lives of DOC to the end of pregnancy
* Women who have exposure to methotrexate or an oral retinoid
* Retrospective enrollment after the outcome of pregnancy is known (ie, the pregnancy has ended prior to enrollment)
* Results of a diagnostic test are positive for an MCM prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate an MCM

Cohort 3: Non-disease unexposed comparator cohort

* Pregnant women who have enrolled in this cohort study with a previous pregnancy
* Women who have had exposure to deucravacitinib or any other oral TYK2 inhibitor, or any oral JAK inhibitor from within 5 half-lives of DOC to the end of pregnancy
* Retrospective enrollment after the outcome of pregnancy is known (ie, the pregnancy has ended prior to enrollment)
* Results of a diagnostic test are positive for an MCM prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate an MCM
* Women exposed to a known, possible, or suspected human teratogen during pregnancy as confirmed by the OTIS Research Center (see Appendix 3 for list of known, possible, and suspected human teratogens)
* Women who are diagnosed with PsO, or any other autoimmune disease

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include pregnant women participating in the The Organization of Teratology Information Specialists (OTIS) pregnancy registry in the US or Canada
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of major congenital malformations among infants | 1-year post pregnancy outcome

SECONDARY OUTCOMES:
Number of other pregnancy and infant outcomes | 1-year post pregnancy outcome
  Other pregnancy and infant outcomes include:
  * Minor congenital malformations,
  * Small for gestational age
  * Small for age postnatal growth at 1 year of age
  * Serious or opportunistic infections
  * Neonatal hospitalization
  * Infant deaths
  * Neonatal deaths
  * Perinatal deaths
  * Spontaneous abortions
  * Stillbirths
  * Elective terminations/abortions
  * Preterm deliveries
  * Preeclampsia/eclampsia
  * Gestational hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts